CLINICAL TRIAL: NCT04470843
Title: Impact of Acetazolamide in Reducing Referred Postoperative Pain After Robotic Assisted Laparoscopic Prostatectomy
Brief Title: Impact of Acetazolamide in Reducing Referred Postoperative Pain
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Scott Johnson, Assistant Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRO00031299
Record Dates: First submitted 2018-08-27; First posted 2020-07-14 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Prostate Cancer; Men
Keywords: Prostatectomy; Acetazolamide; Postoperative Pain; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms; Multiple Endocrine Neoplasia Type 1; Pain, Postoperative | interventions — Acetazolamide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acetazolamide (Active Comparator): Group 1 (acetazolamide): Patients undergoing RALP with the peri-operative use of one-time 250 mg dose of acetazolamide
  Interventions: Drug: Acetazolamide
- Placebo (Placebo Comparator): Group 2 (placebo): Patients undergoing RALP with the peri-operative use of 10 mL normal saline as placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Acetazolamide — Being that adequate pain control is essential to recovery in the post-operative setting, efforts have been made to address this pain at its root. Prior studies have demonstrated that preoperative administration of acetazolamide decreased post-operative referred pain in the immediate post-surgical period.
  Arms: Acetazolamide
Other: Placebo — Group 2 (placebo): Patients undergoing RALP with the peri-operative use of 10 mL normal saline as placebo.
  Arms: Placebo

SUMMARY:
Robotic assisted laparoscopic prostatectomy (RALP) is the standard treatment for prostate cancer, due to the benefits of decreased blood loss and length of stay.The procedure involves removing a man's prostate using a minimally invasive robotic approach under the guidance of a surgeon. In order to gain sufficient access, carbon dioxide (CO2) is used to fill the surgical space in a process termed insufflation. Carbon dioxide is a mainstay in laparoscopic procedures because it is cost-effective, noncombustible and readily excreted via the respiratory system in healthy patients.

Insufflation with CO2, however, has been linked to post-operative referred pain secondary to peritoneal acidosis.This acidosis is suspected to be due to the formation of carbonic acid from the CO2 insufflation.Peritoneal acidosis, and its associated post-operative referred pain, may not be adequately treated with the current standard pain control regimen.

ELIGIBILITY:
Inclusion Criteria:

• Male patients ≥18 years of age undergoing robotic-assisted prostatectomy

Exclusion Criteria:

* Patients with renal insufficiency with serum creatinine >2.0 mg/dl
* Patients with renal transplant
* Patients with pre-existing metabolic acidosis
* Patients with chronic obstructive pulmonary disease
* Patients with hepatic disease
* Patients with central nervous system disorders
* Patients with hematological disease history
* Patients with pre-existing electrolyte abnormalities
* Patients with hypovolemia
* Patients with lithium or diuretic usage
* Patients with sulfonamides allergy
* Patients with American Society of Anesthesiologists physical status 4 or 5

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Males having a robotic-assisted prostatectomy
Enrollment: 33 (Actual)
Dates: Start 2018-08-22 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) 10-cm lines anchored at the ends by words that define the bounds of various pain dimensions. The patient is asked to place a vertical mark on the scale to indicate the level of intensity of his pain. | 24 hours
  The primary outcome to be assessed is the absolute change in VAS score both in general and at the shoulder tip. This will be measured as the difference between the VAS score obtained pre-operatively, when first responsive after surgery in the post anesthesia care unit (PACU), immediately prior to leaving PACU, and throughout the hospital stay per standard of care.
  Δ VAS = Postoperative VAS - Preoperative VAS VAS is a testing technique for measuring subjective or behavioral phenomena (as pain or dietary consumption) in which a subject selects from a gradient of alternatives (as from "no pain" to "worst imaginable pain" or from "every day" to "never") arranged in linear fashion -abbreviation VAS

CONTACTS AND LOCATIONS:
Overall Officials: Scott Johnson, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Memorial Lutheran Hospital, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No